CLINICAL TRIAL: NCT01967108
Title: The Effect of Post Extubation Chest Physiotherapy on Respiratory Complications and Weaning Failure in Critically Ill Patients
Brief Title: Post Extubation Chest Physiotherapy in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0346-13-RMB CTIL
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2014-02

CONDITIONS: Weaning From Mechanical Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- chest physiotherapy (Experimental): chest physiotherapy in patient's bed, including deep breathing, directed cough, arm movment and more.
  Interventions: Other: chest physiotherapy
- control group (No Intervention): This patients will not recive chest physiotherapy after extubation, unless developing respiratory deterioration

INTERVENTIONS:
Other: chest physiotherapy — chest physiotherapy, up to one hour from extubation, in ICU patients
  Arms: chest physiotherapy

SUMMARY:
The purpose of this study is to examine the efficacy of chest physiotheray treatment in preventing pulmonary complications and weaning faliure, in extubated critically ill patients.

ELIGIBILITY:
Inclusion Criteria:ICU patients, over 18 years' old, mechanical ventilated over 24 hours, candidates for extubation -

Exclusion Criteria: Mental conditions, retardation, dementia, pregnancy, re-intubated patients

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
re-intubation | 48 hours
  re-intubation up to 48 hours post extubation will be considered a weaning failure

SECONDARY OUTCOMES:
oxygen saturation decrease | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Enbar Foox, B.PT, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Intensive Care Unit, Rambam Health Care Campus, Haifa, Israel